CLINICAL TRIAL: NCT04675242
Title: Multi-Center, Randomized, Double-Masked, Placebo-Controlled, Phase 2b Study Evaluating the Safety and Efficacy of NCX 4251 Ophthalmic Suspension, 0.1% QD for the Treatment of Acute Exacerbations of Blepharitis (Mississippi)
Brief Title: Study Evaluating the Safety and Efficacy of NCX 4251 Ophthalmic Suspension for the Treatment of Blepharitis
Acronym: Mississippi
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nicox Ophthalmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCX-4251-02
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Results first posted 2022-12-14 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Blepharitis
MeSH Terms: conditions — Blepharitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NCX 4251 (Experimental): NCX 4251 Ophthalmic Suspension
  Interventions: Drug: NCX 4251
- Placebo (Placebo Comparator): Vehicle of NCX 4251 Ophthalmic Suspension
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NCX 4251 — NCX 4251 Ophthalmic Suspension, 0.1% dosed once daily
  Arms: NCX 4251
Drug: Placebo — Vehicle of NCX 4251 Ophthalmic Suspension dosed once daily
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-masked, placebo-controlled, Phase 2b trial evaluating the safety and efficacy of NCX 4251 (fluticasone propionate nanocrystal) Ophthalmic Suspension 0.1% QD for the treatment of acute exacerbations of blepharitis.

ELIGIBILITY:
Inclusion Criteria:

* documented history of blepharitis and meet qualifying criteria for an acute exacerbation of blepharitis in both eyes at Screening and Baseline/Day 1 Visits
* have a qualifying best-corrected visual acuity

Exclusion Criteria:

* abnormality of the eyelids or lashes (other than blepharitis), or previous eyelid surgery
* IOP > 21 mmHg at Screening or Baseline/Day 1 Visits
* use of steroids in the past 30 days or retinoids in the past 12 months
* uncontrolled systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicox Ophthalmics, Study Director — Nicox Ophthalmics, Inc.
Locations (1):
- Eye Research Foundation, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: eyecare practictioners' practices
Pre-assignment Details: 7 to 14 day screening period
Units Other Than Participants: study eye
Period: Overall Study
Arm/Group | NCX 4251 | Placebo
Started | 111; 111 study eye | 113; 113 study eye
Completed | 109; 109 study eye | 112; 112 study eye
Not Completed | 2; 2 study eye | 1; 1 study eye

BASELINE CHARACTERISTICS:
Population: Study Eye
Groups:
- Total: Total of all reporting groups
Arm/Group | NCX 4251 | Placebo | Total
Number analyzed (Participants) | 111 | 113 | 224
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 50 | 113
  >=65 years | 48 | 63 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (13.75) | 63.2 (14.31) | 62.3 (14.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 67 | 142
  Male | 36 | 46 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 106 | 105 | 211
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 21 | 47
  White | 84 | 87 | 171
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 111 | 113 | 224
Composite Score of Eyelid Margin Redness + Eyelid Debris + Eyelid Discomfort in the study eye [Mean (Full Range); unit: units on a scale for study eyes] — Composite (sum) score of Eyelid Margin Redness (0=none to 3=severe), Eyelid Debris (0=none to 3=severe), and Eyelid Discomfort (0=none to 3=severe) in the study eye
  units on a scale for study eyes | 4.6 [3 to 8] | 4.7 [3 to 7] | 4.7 [3 to 7]
Eye Dryness [Mean (Full Range); unit: units on a scale for study eyes] — visual analog scale (0=no discomfort to 100=maximal discomfort)
  units on a scale for study eyes | 59.1 [4 to 99] | 57.5 [0 to 99] | 58.3 [0 to 99]
Inferior Cornea Staining Score [Mean (Full Range); unit: units on a scale for study eyes] — Fluorescein staining scale (0=none to 4=severe)
  units on a scale for study eyes | 1.70 [0 to 3.5] | 1.69 [0 to 4.0] | 1.70 [0 to 4.0]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Study Eyes With Complete Cure (Score 0) of Blepharitis Signs and Symptoms at Day 15
Description: Percentage of study eyes with Complete Cure (Score 0) in each of the following: Eyelid Margin Redness (0-none, 1-mild, 2-moderate, 3-severe), Eyelid Debris (0-none, 1-mild, 2-moderate, 3-severe), and Eyelid Discomfort (0-none, 1-mild, 2-moderate, 3-severe) at the Day 15 Visit
Time Frame: Day 15 Visit
Population: Intent to treat (for study eyes with data for all 3 scales at the Baseline and Day 15 Visit)
Measure: Count of Units; unit: study eyes
Units Other Than Participants: study eyes
Arm/Group | NCX 4251 | Placebo
Number analyzed (Participants) | 109 | 111
Number analyzed (study eyes) | 109 | 111
study eyes | 4 | 2
Statistical Analysis 1: Comparison: NCX 4251 vs Placebo; Difference in the proportion of study eyes with complete cure; Test type: Superiority; p = 0.4434, Fisher Exact; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-11.5 to 15.3]

2. Secondary Outcome: Mean Change From Baseline to Day 15 in Study Eye Eye Dryness Symptoms
Description: Mean change from baseline in the eye dryness symptoms using a visual analogue scale (0 = no discomfort to 100 = maximal discomfort) at the Day 15 Visit
Time Frame: Day 15 Visit
Population: intent to treat (in study eyes with data at Baseline and Day 15 Visit)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: study eyes
Arm/Group | NCX 4251 | Placebo
Number analyzed (Participants) | 109 | 112
Number analyzed (study eyes) | 109 | 112
units on a scale | -16.4 [-20.7 to -12.0] | -12.5 [-16.5 to -8.5]
Statistical Analysis 1: Comparison: NCX 4251 vs Placebo; Difference in the change from baseline between treatment groups; Test type: Superiority; p = 0.2105, ANCOVA; adjusted for baseline eye dryness VAS score; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-9.5 to 2.1]

3. Secondary Outcome: Mean Change From Baseline to Day 15 in Study Eye Eye Dryness Sign (Fluorescein Staining of the Inferior Cornea)
Description: Mean change from baseline in study eye fluorescein staining score (score of 0=none, 1=trace, 2=mild, 3=moderate, 4=severe) of the inferior cornea at the Day 15 Visit
Time Frame: Day 15 Visit
Population: intent to treat (for study eyes with data at Baseline and Day 15)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: study eyes
Arm/Group | NCX 4251 | Placebo
Number analyzed (Participants) | 109 | 112
Number analyzed (study eyes) | 109 | 112
units on a scale | -0.18 [-0.34 to -0.02] | -0.13 [-0.26 to 0.01]
Statistical Analysis 1: Comparison: NCX 4251 vs Placebo; Difference in the mean change from baseline; Test type: Superiority; p = 0.5936, ANCOVA; adjusted for baseline eye dryness VAS score; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.1]

4. Secondary Outcome: Treatment-emergent Adverse Events
Description: Number of participants with treatment-emergent adverse events (an adverse event that occurred on or after treatment with the intervention was initiated)
Time Frame: 29 days
Population: Safety population (all randomized subjects who received at least one dose of the intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | NCX 4251 | Placebo
Number analyzed (Participants) | 111 | 113
Participants | 12 | 17

ADVERSE EVENTS:
Time Frame: 29 days
Arm/Group | NCX 4251 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/113
Other Adverse Events (participants affected / at risk) | 12/111 | 20/113
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NCX 4251 (N=111) | Placebo (N=113)
Visual acuity reduced (Eye disorders) | 1 (1) | 2 (2)
Eye pruritus (Eye disorders) | 1 (1) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (1) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Eyelid irritation (Eye disorders) | 0 (0) | 1 (1)
Eyelids pruritus (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Instillation site pain (General disorders) | 1 (1) | 5 (5)
Instillation site oedema (General disorders) | 0 (0) | 1 (1)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Splinter (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT04675242/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT04675242/SAP_001.pdf